CLINICAL TRIAL: NCT02702258
Title: Mindfulness-Based Blood Pressure Reduction (MB-BP) Stage 1 Single Arm Trial: Acceptability and Feasibility Study; Additionally Exploring the Preliminary Effects on Self-Regulation Targets, Including Self Awareness, Emotion Regulation and Attention Control
Brief Title: Mindfulness-Based Blood Pressure Reduction (MB-BP) Intervention Development - Stage 1 Single Arm Trial
Acronym: MB-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Eric Loucks, Assistant Professor, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1412001171-1; 1UH2AT009145-01 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Prehypertension; Hypertension
Keywords: mindfulness; blood pressure; hypertension; prehypertension
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MB-BP (Experimental): This is the primary intervention tested in this single arm trial.
  Interventions: Behavioral: MB-BP

INTERVENTIONS:
Behavioral: MB-BP — MB-BP (Mindfulness-Based Blood Pressure Reduction) customizes Mindfulness-Based Stress Reduction (MBSR) to participants with prehypertension/hypertension. MB-BP will consist of nine 2.5-hour weekly group sessions and an 7.5-hour one-day session. Some of the unique areas of MB-BP are education on hypertension risk factors, hypertension health effects, and specific mindfulness modules focused on awareness of blood pressure determinants such as diet, physical activity, antihypertensive medication adherence, alcohol consumption, and stress reactivity. Students learn a range of mindfulness skills including body scan exercises, meditation and yoga. Homework consists of practicing skills for ≥45 min/day, 6 days/week.

SUMMARY:
Specific aims are:

1. To outline and evaluate key active elements of the Mindfulness-Based Blood Pressure Reduction (MB-BP) intervention. This aim will be achieved using (a) focus groups of participants undergoing the MB-BP intervention, (b) discussion with experts (including cardiologists, epidemiologists, mindfulness experts, mindfulness intervention instructors) prior to, and following pilot testing of MBHT in participants, and (c) clinical judgment of the investigators performing the intervention.
2. To evaluate impacts of MB-BP on target engagement (pre-post change in effect size) and longevity of target engagement (follow-up time-points). Follow-up time periods include 10 weeks, 6 months and 1 year.

This study is a prospective single-arm trial during the intervention development phase. Following this phase, after the intervention has been further developed, a subsequent study (with a different clinicaltrials.gov identification #) will utilize a randomized control trial design to further evaluate causation and effect size.

DETAILED DESCRIPTION:
Mindfulness interventions customized for prehypertensive/hypertensive patients have never been investigated. Until methodologically rigorous studies to evaluate customized interventions for hypertension are performed, we will not know if the observed preliminary effects of general mindfulness interventions on blood pressure reduction could be much more effective with a tailored approach. Consequently, we propose to conduct a behavioral intervention study to evaluate whether Mindfulness-Based Stress Reduction (MBSR) customized to prehypertensive and hypertensive patients has the potential to provide clinically relevant reductions in blood pressure. This customized intervention is called Mindfulness-Based Blood Pressure Reduction (MB-BP). This study follows the NIH Stage Model for Behavioral Intervention Development, where targets likely proximally affected by the intervention are identified, that should also have effect on the longer-term outcomes (e.g. blood pressure, mortality). The selected targets, consistent with theoretical frameworks and early evidence how mindfulness interventions could influence mental and physical health outcomes, are measures of self-regulation including (1) attention control (specifically the Sustained Attention Response Task), (2) emotion regulation (specifically the Difficulty in Emotion Regulation Scale), and (3) self-awareness (specifically the Multidimensional Assessment of Interoceptive Awareness). Based on the degree of target engagement, MB-BP can be further customized to better engage with the targets as needed. The grant funding this study is performing a concurrent systematic review of impacts of mindfulness interventions on self-regulation outcomes. Based on the findings from the systematic review, other self-regulation measures will be explored as secondary outcomes.

Specific aims are:

1. To outline and evaluate key active elements of MB-BP. This aim will be achieved using (a) focus groups of participants undergoing the MB-BP intervention, (b) discussion with experts (including cardiologists, epidemiologists, mindfulness experts, mindfulness intervention instructors) prior to, and following pilot testing of MBHT in participants, and (c) clinical judgment of the investigators performing the intervention.
2. To evaluate impacts of MB-BP on target engagement (pre-post change in effect size) and longevity of target engagement (follow-up time-points). Follow-up time periods include 10 weeks, 6 months and 1 year.

This study is a prospective single-arm trial during the intervention development phase. Following this phase, after the intervention has been further developed, a subsequent study (with a different clinicaltrials.gov ID #) will utilize a randomized control trial design to further evaluate causation and effect size.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension/prehypertension (≥120 mmHg systolic, ≥80 mmHg diastolic pressure or taking antihypertensive medication).
* Able to speak, read, and write in English.
* All adults (≥18 years of age), genders and racial/ethnic groups are eligible to be included.

Exclusion Criteria:

* Current regular meditation practice (>once/week)
* Serious medical illness precluding regular class attendance
* Current substance abuse, suicidal ideation or eating disorder
* History of bipolar or psychotic disorders or self-injurious behaviors. These participants are excluded because they may disrupt group participation, require additional or specialized treatment, or are already participating in practices similar to the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Sustained Attention to Response Task | 1 year follow-up
  The Sustained Attention Test is a computer-based task designed to measure a person's ability to withhold responses to infrequent and unpredictable stimuli during a period of rapid and rhythmic responding to frequent stimuli.
Difficulties in Emotion Regulation Scale | 1 year follow-up
  This is a brief, 36-item, self-report questionnaire designed to assess multiple aspects of emotion dysregulation.
Multidimensional Assessment of Interoceptive Awareness | 1 year follow-up
  This measure assesses interoceptive awareness across multiple domains such as awareness of body sensations, trusting body sensations, and mind-body integration.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Loucks, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Individuals interested in utilizing data are welcome to contact the principal investigator with a data analysis proposal.

REFERENCES:
- [Result] Loucks EB, Nardi WR, Gutman R, Kronish IM, Saadeh FB, Li Y, Wentz AE, Webb J, Vago DR, Harrison A, Britton WB. Mindfulness-Based Blood Pressure Reduction (MB-BP): Stage 1 single-arm clinical trial. PLoS One. 2019 Nov 27;14(11):e0223095. doi: 10.1371/journal.pone.0223095. eCollection 2019. PMID 31774807
- See also: Mindfulness-Based Blood Pressure Reduction (MB-BP): Stage 1 single-arm clinical trial — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0223095

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT02702258/Prot_SAP_ICF_000.pdf